CLINICAL TRIAL: NCT02337101
Title: Early Intervention Programme for Impairing Post-concussional Symptoms in Adolescents and Young Adults: Randomised Trial
Brief Title: Early Intervention Programme for Young Patients (Aged 15 - 30 Years) With Symptoms Following Concussion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Central Denmark Region (Other); Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18122014
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-01

CONDITIONS: Brain Concussion; Post-Concussion Syndrome
Keywords: Brain concussion; Mild Traumatic Brain Injury; Post-concussion symptoms; Therapy; Randomised controlled trial; Cognitive assessment
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): Clinical psychiatric and neurological assessment. Information and advice.
  Interventions: Other: Enhanced Usual Care (EUC)
- EUC + Early intervention programme (Experimental): Clinical psychiatric and neurological assessment. Information and advice. Individually targeted treatment programme.
  Interventions: Behavioral: EUC + Early intervention programme

INTERVENTIONS:
Other: Enhanced Usual Care (EUC) — All patients will have a brief clinical psychiatric and neurological assessment in order to determine eligibility, and will be provided with information and advice about typical post-concussional symptoms, the typical recovery process and the use of pain medication.
  Arms: Enhanced Usual Care (EUC)
Behavioral: EUC + Early intervention programme — All patients will have a brief clinical psychiatric and neurological assessment in order to determine eligibility, and will be provided with information and advice about typical post-concussional symptoms, the typical recovery process and the use of pain medication.
  The early intervention programme will be interdisciplinary and will mainly be provided by an occupational therapist and a physiotherapist under supervision of a neuropsychologist. It will be based on psychoeducation and principles from Cognitive Behavioral Therapy and Graded Exercise Therapy and targeted to patients' individual goals.
  Patients will receive 8 weekly treatment sessions (3 group based and 5 individual sessions). Intervention will start approximately 4-5 months after the concussion.
  Arms: EUC + Early intervention programme

SUMMARY:
Background:

Five - 15 % of patients with concussion continue to experience impairing physical, cognitive and emotional symptoms longer than 3 months post-injury. Currently, no standardised treatment is available for patients with persistent post-concussional symptoms (PCS) and systematic treatment studies remain limited.

Aim:

1. to develop an early intervention programme based on principles from cognitive-behavioural therapy and graded exercise for young patients with PCS lasting more than 3 months, and
2. to evaluate the efficacy of this intervention on PCS in a randomised, controlled trial.

Methods:

Patients aged 15 - 30 years diagnosed with concussion at hospitals in Central Denmark Region will be screened for persistent symptoms two months post-injury. Those with impairing symptoms will be invited to participate in a randomised controlled trial comparing the early intervention programme with enhanced usual care. We expect to include 120 patients from 2015-2016. Treatment will be interdisciplinary and will begin approximately 3 - 5 months after concussion. All patients will complete self-report measures at baseline and 3, 6 and 15 months after randomisation. The primary outcome is severity of PCS.

DETAILED DESCRIPTION:
Background Concussion is an important public health concern. Debilitating and persistent post-concussional symptoms are associated with considerable long-term sickness and markedly reduced health-related quality of life in industrialized countries. In Denmark, approximately 25000 people are diagnosed with concussion each year. Although complete resolution of typical post-concussional symptoms such as headaches, dizziness and fatigue normally occur within the first days or weeks after a concussion, a significant proportion corresponding to five to15 % of patients continue to experience symptoms longer than 3 months post-injury. These patients are at risk of long-term sickness, reduced health-related quality of life as well as permanently reduced working ability, which is particularly disastrous for adolescents and young adults. Currently, no standardised treatment is available for patients with persistent post-concussional symptoms.

The aetiology of persistent post-concussional symptoms is only partly elicited, and no consensus exists whether post-concussional symptoms constitute a true syndrome linked to neurobiological disturbances caused by accident or head trauma. Nevertheless, the term post-concussional syndrome is widely used to describe a set of persistent somatic and emotional symptoms often observed in concussed individuals. We use the abbreviation 'PCS' as a purely descriptive term for post-concussional symptoms. The literature suggest, that PCS are best understood in a complex, multifactorial model, where both biological and psychological factors contribute to persistent symptoms and associated disability. Moreover, PCS overlap considerably with symptoms of other trauma-related conditions such as whiplash-associated disorders and post-traumatic stress disorder. On this background, a number of trials have tested the effect of various psychosocial interventions, including cognitive behavioural therapy (CBT), on persistent PCS. Although preliminary, there is some promising evidence that treatment based on the cognitive-behavioural model may be effective in treating PCS and prevent permanent suffering and disability.

Some of the cognitive - behavioural mechanisms that have been found to play an important role in the maintenance of PCS are unhelpful illness perceptions, maladaptive coping strategies and all-or-nothing behaviour. The all-or-nothing behaviour refers to a behavioural response, where patients overdo things when they believe symptoms are abating and then spend prolonged periods recovering when symptoms reappear. Other patients report a gradual restriction of activity over time, because they fear worsening of symptoms. A promising avenue for treatment seems to be focusing on making sustainable, gradual increases in levels of activity (in intensity and / or duration) over time, and to avoid extreme oscillations. This is often referred to as Graded Exercise Therapy (GET), a treatment that can effectively reduce impairment and suffering in chronic fatigue and persistent pain and that can be provided by physiotherapists and hence delivered in a primary care or municipality setting.

Currently, systematic studies of psychosocial interventions for patients with persistent PCS remain limited. A recent review concludes that more rigorous, large-scale randomised controlled trials (RCT) evaluating the effectiveness of CBT for persistent PCS are needed.

Aim:

1. to develop an early intervention programme based on CBT and GET principles for young patients aged 15 - 30 years with PCS lasting more than three months, and
2. to evaluate the efficacy of this intervention programme on PCS in a RCT.

Hypotheses Primary hypothesis Patients in the early intervention group will 6 months after randomisation report a statistically and clinically significantly greater reduction of post-concussional symptoms compared to patients who receive enhanced usual care.

Secondary hypotheses

1. Patients in the early intervention group will 6 months after randomisation report a statistically and clinically significantly higher health related quality of life and overall daily functioning compared to patients who receive enhanced usual care.
2. Patients in the early intervention group will during the 12 months after treatment have less consumption of health care (based on register-data) and less illness-related absence from school or work (based on self-reported data) compared to patients, who receive enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Concussion caused by a head trauma according to the diagnostic criteria recommended by the Danish Consensus Report on Commotio Cerebri 5 within the last 2 - 6 months. The criteria is based on the diagnostic criteria recommended by the WHO Task Force 1, but with the amendment, that there must have been a direct contact between the head and an object in order to rule out acceleration - deceleration traumas.
2. Age between 15 and 30 years at the time of the head trauma.
3. Able to understand, speak and read Danish.
4. A score of 20 or more on the Rivermead Post Concussion Symptoms Questionnaire (RPQ).

Exclusion Criteria:

1. Objective neurological findings from neurological examination and / or acute trauma CT scan, indicating neurological disease or brain damage.
2. Previous concussion leading to persistent post-concussional symptoms within the last two years.
3. Severe misuse of alcohol, prescription drugs and / or illegal drugs.
4. Multiorgan Bodily Distress Syndrome (multiple somatic symptoms from various body sites and organ systems not related to the accident).
5. Psychiatric morbidity (Bipolar Disorder, severe Attention Deficit Hyperactivity Disorder, autism, psychotic disorder (life time)), or other psychiatric illness that impedes participation in the treatment.
6. Severe neurological disease and / or other medical disease that impedes participation in the treatment programme.
7. Significant learning and / or reading difficulties or mental retardation.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Severity of PCS measured by the Rivermead Post-concussion Symptoms Questionnaire (RPQ) | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
  Self-rated post-concussion symptoms

SECONDARY OUTCOMES:
Quality of life and overall functioning measured by Quality of Life After Brain Injury - Overall Scale (QOLIBRI) and Short Form health status questionnaire from the medical outcome status (SF-36). | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
Subjective improvement measured by Patient Global Impression of Change (PGIC) | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
Somatisation measured by Bodily Distress Syndrome Checklist (BDS checklist) | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
Anxiety and depression severity measured by a subscale (SCL-8) of Symptom Check List, 90 items (SCL-90). | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint)and 15 months after baseline.
Health Anxiety measured by Whitely-8 index | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
Consumption of health care (extracted from Danish national registers) and degree of illness related absence from school or work (self-reported). | 15 months after baseline (i.e. after clinical assessment)
Self-reported cognitive functioning measured by Behavior Rating Inventory of Executive Function (BRIEF) | At baseline (i.e. at clinical assessment) and 6 months after baseline (primary endpoint).
Change in illness related cognitions measured by The Brief Illness Perception Questionnaire (B-IPQ) | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
  Process measure
Change in illness-related behaviours measured by the Behavioural Responses to Illness Questionnaire - short form (BRIQ - short form) | At baseline (i.e. at clinical assessment) and 3,6 and 15 months after baseline.
  Process measure
Change in perceived stress measured by Perceived Stress Scale (PSS) | At baseline (i.e. at clinical assessment) and 3,6 (primary endpoint) and 15 months after baseline.
  Process measure

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schröder, MD, PhD, Principal Investigator — Aarhus University Hospital; Charlotte U Rask, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Thastum MM, Rask CU, Naess-Schmidt ET, Tuborgh A, Jensen JS, Svendsen SW, Nielsen JF, Schroder A. Novel interdisciplinary intervention, GAIN, vs. enhanced usual care to reduce high levels of post-concussion symptoms in adolescents and young adults 2-6 months post-injury: A randomised trial. EClinicalMedicine. 2019 Dec 16;17:100214. doi: 10.1016/j.eclinm.2019.11.007. eCollection 2019 Dec. PMID 31891145
- See also: Homepage for the Research Clinic for Functional Disorders, Aarhus University Hospital — http://www.functionaldisorders.dk